CLINICAL TRIAL: NCT01293266
Title: Effect of Propofol and Sevoflurane on Base Excess, pH and Lactate in Pediatric Heart Catheterisation
Brief Title: Effect of Propofol and Sevoflurane on Lactate During Anesthesia for Pediatric Heart Catheterisation
Acronym: PRISCATHLAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Department of Anaesthesiology and Intensive Care Medicine, University Hospital Schleswig-Holstein, Campus Kiel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Fudickar2
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-02

CONDITIONS: Metabolic Acidosis
Keywords: Propofol; Metabolic Acidosis; Pediatric Cardiology; Anesthesia
MeSH Terms: conditions — Acidosis | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): Anesthesia is changed from Sevoflurane to Propofol after obtaining baseline blood gas analysis from the heart catheterisation sheath.
  Interventions: Drug: Propofol
- Sevoflurane (No Intervention): Sevoflurane anesthesia is maintained after obtaining a baseline blood gas analysis.

INTERVENTIONS:
Drug: Propofol — Anesthesia is switched from sevoflurane to propofol after obtaining a baseline blood gas analysis.
  Other Names: Disoprivan
  Arms: Propofol

SUMMARY:
Propofol is routinely used for general anesthesia during pediatric heart catheterisation. Propofol infusion syndrome (PRIS) is a rare, but often fatal complication mainly defined by bradycardia with progress to asystolia during propofol infusion. Metabolic acidosis is regarded as an early warning sign of PRIS. In this study the effect of propofol and sevoflurane on serum base excess, pH and lactate are examined during pediatric heart catheterisation.

DETAILED DESCRIPTION:
In this prospective randomised study 40 children are anesthetised for pediatric heart catheterisation with propofol (N = 22) or sevoflurane (N = 18) with ethic committee approval. Base excess, pH and lactate were measured by blood gas analysis at the beginning, during and at the end of the procedure. Changes relative to baseline were analysed by paired t-Test with correction for multiple testing. The study was powered to detect a difference of 1.5 mmol/l for base excess and lactate.

ELIGIBILITY:
Inclusion Criteria:

* Indication for heart catheterization under general anesthesia

Exclusion Criteria:

* Participation in another study
* Preexisting metabolic acidosis
* Contraindication against Propofol

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Serum Lactate | 4 hours
  Serum lactate is measured during application of propofol and sevoflurane to examine the effect on metabolic acidosis.

SECONDARY OUTCOMES:
pH and base excess | Hours
  pH and base excess are measured during application of Propofol and Sevoflurane to examine the effect on acid-base balance

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Bein, Prof. Dr., Study Director — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany